CLINICAL TRIAL: NCT05958264
Title: Evaluation of Sublingual Microcirculation Using Sidestream Dark-Field Imaging in Children with Type 1 Diabetes Mellitus with Favorable Treatment Outcomes.
Brief Title: Sublingual Microcirculation in Children with Compensated T1D Using the SDF Method
Status: Completed | Type: Observational
Sponsor: Vlasta Krausová (Other)
Responsible Party: Sponsor-Investigator, Vlasta Krausová, Principal Investigator, Masarykova Nemocnice v Usti nad Labem, Krajska Zdravotni a.s.
Organization: Masarykova Nemocnice v Usti nad Labem, Krajska Zdravotni a.s. (Other)
Other Study IDs: 310/1
Record Dates: First submitted 2023-06-28; First posted 2023-07-24 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Type1diabetes
Keywords: Microcirculation; Children; Type1diabetes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Children of younger school age: 10 children of younger school age aged 6-10,9 years with T1D.
- Children in puberty: 10 children in puberty aged 11-14,9 years with T1D
- Postpubertal adolescents: 10 postpubertal adolescents aged 15-18,9 years with T1D

SUMMARY:
The main goal of the study is to describe the sublingual microcirculation of children with type 1 diabetes mellitus (T1D) with stable and satisfactory treatment of the disease and to compare it with previously measured parameters of healthy children, NCT05324228.

DETAILED DESCRIPTION:
After recording the basic anthropometric parameters, pressure and pulse, each child who meets the inclusion criteria will have their microcirculation measured using a Sidestream Dark-Field (SDF) probe placed sublingually by one examiner using the SDF method. The measurement will be performed in supine position in a disease-free period, with normal diets, at least 2 hours after the last meal, for girls outside the menses period. Premedication or analgesia will not be used. A total of 3 video clips will be recorded from different parts of the sublingual area with a minimum length of 20 seconds in a row, unless the child needs a short break between measurements. The recorded videos will then be processed offline by one evaluator who is trained and experienced in microcirculation evaluation, three best and most stable parts of each video clip will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes mellitus
* informed consent of parents

Exclusion Criteria:

* acute infection
* period of metabolic decompensation and 14 days after it

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will include 40 children with T1D. Of these, 10 pre-school children (3-5.9 years), 10 younger school children (6-10.9 years), 10 children in puberty(11-14.9 years) and 10 post-puberty adolescents will be included (15-18.9 years).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Determination of Total Vascular Density of sublingual microcirculation of children with T1D | baseline
  Total length of vessels divided by total surface of area
Determination of Microvascular Flow Index (MFI) of sublingual microcirculation of children with T1D | baseline
  The image is divided into four quadrants and the predominant type of flow (absent = 0, intermittent = 1, sluggish = 2, normal = 3, and hyperdynamic = 4) is assessed in each quadrant. The MFI score represents the averaged values of the four. A 20 μm cut-off is used to separate small vessels (mostly capillaries) from large vessels (mostly venules).
Determination of Small Vessel Density of sublingual microcirculation of children with T1D | baseline
  Total length of small vessels divided by total surface of area. A 20 μm cut-off is used to separate small vessels (mostly capillaries) from large vessels (mostly venules).
Determination of Proportion of Perfused Vessels (all) of sublingual microcirculation of children with T1D | baselina
  The proportion of perfused vessels (PPV [%]) can be calculated as follows: 100 × (total number of vessels - [no flow + intermittent flow])/total number of vessels.
Determination of Proportion of Perfused Small Vessels (PPSV) of sublingual microcirculation of children with T1D | baseline
  The proportion of perfused small vessels (PPSV [%]) can be calculated as follows: 100 × (total number of small vessels - [no flow + intermittent flow])/total number of small vessels.
  A 20 μm cut-off is used to separate small vessels (mostly capillaries) from large vessels (mostly venules).
Determination of Perfused Vessel Density (PVD) of sublingual microcirculation of children with T1D | baseline
  Total length of vessels - (no flow + intermittent flow) divided by total surface of area
Determination of Perfused Small Vessel Density (PSVD) of sublingual microcirculation of children with T1D | baseline
  Total length of small vessels - (small vessels with no flow + intermittent flow) divided by total surface of area. A 20 μm cut-off is used to separate small vessels (mostly capillaries) from large vessels (mostly venules).
Determination of DeBacker Score of sublingual microcirculation of children | baseline
  In this score, three equidistant horizontal and three equidistant vertical lines are drawn on the screen. Vessel density can be calculated as the number of vessels crossing the lines divided by the total length of the lines. Higher number means better microcirculation.

SECONDARY OUTCOMES:
Differences in Total Vascular Density of sublingual microcirculation in different age and gender categories in children with T1D | baseline
  Comparison in children aged 6-10,9; 11-14,9; and 15-18,9 years and males vs. females.
Differences in Microvascular Flow Index (MFI) of sublingual microcirculation in different age and gender categories in children with T1D | baseline
  Comparison in children aged 6-10,9; 11-14,9; and 15-18,9 years and males vs. females.
Differences in Small Vessel Density of sublingual microcirculation in different age and gender categories in children with T1D | baseline
  Comparison in children aged 6-10,9; 11-14,9; and 15-18,9 years and males vs. females.
Differences Proportion of Perfused Vessels (all) of sublingual microcirculation in different age and gender categories in children with T1D | baseline
  Comparison in children aged 6-10,9; 11-14,9; and 15-18,9 years and males vs. females.
Differences in Proportion of Perfused Small Vessels (PPSV) of sublingual microcirculation in different age and gender categories in children with T1D | baseline
  Comparison in children aged 6-10,9; 11-14,9; and 15-18,9 years and males vs. females.
Differences in Perfused Vessel Density (PVD) of sublingual microcirculation in different age and gender categories in children with T1D | baseline
  Comparison in children aged 6-10,9; 11-14,9; and 15-18,9 years and males vs. females.
Differences in Perfused Small Vessel Density (PSVD) of sublingual microcirculation in different age and gender categories in children with T1D | baseline
  Comparison in children aged 6-10,9; 11-14,9; and 15-18,9 years and males vs. females.
Differences in DeBacker Score of sublingual microcirculation in different age and gender categories in children with T1D | baseline
  Comparison in children aged 6-10,9; 11-14,9; and 15-18,9 years and males vs. females. Higher number means better microcirculation.
Correlation of Total Vascular Density of sublingual microcirculation with parameters of diabetic compenzation | baseline
  Comparison of parametes in children with good and bad compenzation of T1D
Correlation of Microvascular Flow Index (MFI) of sublingual microcirculation with parameters of diabetic compenzation | baseline
  Comparison of parametes in children with good and bad compenzation of T1D
Correlation of Small Vessel Density of sublingual microcirculation with parameters of diabetic compenzation | baseline
  Comparison of parametes in children with good and bad compenzation of T1D
Correlation of Proportion of Perfused Vessels (all) of sublingual microcirculation with parameters of diabetic compenzation | baseline
  Comparison of parametes in children with good and bad compenzation of T1D
Correlation of Proportion of Perfused Small Vessels (PPSV) of sublingual microcirculation with parameters of diabetic compenzation | baseline
  Comparison of parametes in children with good and bad compenzation of T1D
Correlation of Perfused Vessel Density (PVD) of sublingual microcirculation with parameters of diabetic compenzation | baseline
  Comparison of parametes in children with good and bad compenzation of T1D
Correlation of Perfused Small Vessel Density (PSVD) of sublingual microcirculation with parameters of diabetic compenzation | baseline
  Comparison of parametes in children with good and bad compenzation of T1D
Correlation of DeBacker Score of sublingual microcirculation with parameters of diabetic compenzation | baseline
  Comparison of parametes in children with good and bad compenzation of T1D
Differences of Total Vascular Density of sublingual microcirculation with parameters of healthy children in the same age categories | baseline
  Total Vascular Density of sublingual microcirculation of healthy children has been obtained previously within study NCT05324228
Differences of Microvascular Flow Index (MFI) of sublingual microcirculation with parameters of healthy children in the same age categories | baseline
  Microvascular Flow Index (MFI) of sublingual microcirculation of healthy children has been obtained previously within study NCT05324228
Differences of Small Vessel Density of sublingual microcirculation with parameters of healthy children in the same age categories | baseline
  Small Vessel Density of sublingual microcirculation of healthy children has been obtained previously within study NCT05324228
Differences of Proportion of Perfused Vessels (all) of sublingual microcirculation with parameters of healthy children in the same age categories | baseline
  Proportion of Perfused Vessels (all) of sublingual microcirculation of healthy children has been obtained previously within study NCT05324228
Differences of Proportion of Perfused Small Vessels (PPSV) of sublingual microcirculation with parameters of healthy children in the same age categories | baseline
  Proportion of Perfused Small Vessels (PPSV) of sublingual microcirculation of healthy children has been obtained previously within study NCT05324228
Differences of Perfused Vessel Density (PVD) of sublingual microcirculation with parameters of healthy children in the same age categories | baseline
  Perfused Vessel Density (PVD) of sublingual microcirculation of healthy children has been obtained previously within study NCT05324228
Differences of Perfused Small Vessel Density (PSVD) of sublingual microcirculation with parameters of healthy children in the same age categories | baseline
  Perfused Small Vessel Density (PSVD) of sublingual microcirculation of healthy children has been obtained previously within study NCT05324228
Differences of DeBacker Score of sublingual microcirculation with parameters of healthy children in the same age categories | baseline
  DeBacker Score of sublingual microcirculation of healthy children has been obtained previously within study NCT05324228

CONTACTS AND LOCATIONS:
Overall Officials: David Neumann, MD, Ph.D., Study Chair — Hospital in Trutnov
Locations (1):
- Masarykova Nemocnice v Usti nad Labem, Krajska Zdravotni a.s., Ústí nad Labem, Czechia

REFERENCES:
- [Derived] Krausova V, Neumann D, Stichova L, Skvor J, Dostalova V, Dostal P. Alterations of Sublingual Microcirculation in Children With Compensated Type 1 Diabetes Mellitus-An Observational Study. Pediatr Diabetes. 2025 Sep 30;2025:8811411. doi: 10.1155/pedi/8811411. eCollection 2025. PMID 41064468